CLINICAL TRIAL: NCT01947855
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, 4-week Study to Evaluate the Efficacy of Empagliflozin (10 mg and 25 mg Administered Orally Once Daily) in Postprandial Glucose and 24-hour Glucose Variability in Japanese Patients With Type 2 Diabetes Mellitus With Insufficient Glycaemic Control
Brief Title: Post Prandial Glucose (PPG) Study of Empagliflozin in Japanese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.35
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (3):
- Empagliflozin low dose (Experimental): Empagliflozin low dose tablet once daily
  Interventions: Drug: Empagliflozin; Drug: Placebo
- Empagliflozin high dose (Experimental): Empagliflozin high dose tablet once daily
  Interventions: Drug: Placebo; Drug: Empagliflozin
- Placebo (Placebo Comparator): Placebo tablet once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo tablet matching Empagliflozin low dose
  Arms: Empagliflozin high dose
Drug: Empagliflozin — Empagliflozin low dose
  Arms: Empagliflozin low dose
Drug: Placebo — Placebo tablet matching Empagliflozin high dose
  Arms: Placebo
Drug: Placebo — Placebo tablet matching Empagliflozin low dose
  Arms: Placebo
Drug: Empagliflozin — Empagliflozin high dose tablet once daily
  Arms: Empagliflozin high dose
Drug: Placebo — Placebo tablet matching Empagliflozin high dose
  Arms: Empagliflozin low dose

SUMMARY:
To evaluate the efficacy of empagliflozin administered orally once daily in postprandial glucose and 24-hour glycaemic variability compared to placebo given for 4 weeks as mono-therapy in Japanese patients with type 2 diabetes mellitus with insufficient glycaemic control on no antidiabetic treatment.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of type 2 diabetes mellitus prior to informed consent
* Male and female patients on diet and exercise regimen for 12 weeks prior to informed consent who are:

  * drug-naïve, defined as no antidiabetic drugs for at least 12 weeks prior to informed consent or,
  * pre-treated with one oral antidiabetic drug (except sulfonylurea and thiazolidinedione); the present antidiabetic therapy has to be unchanged for at least 12 weeks prior to the informed consent. (Sulfonylurea is permitted as pre-treatment drug only if the dose is equal or less than a half of daily maximum approval dose.)
* Glycosylated haemoglobin (HbA1c) at Visit 1 (screening)

  * for patients without antidiabetic therapy : HbA1c >=7.0 to =<10.0%
  * for patients with one oral antidiabetic drug : HbA1c >=7.0 to =<9.5%

Exclusion criteria:

* Uncontrolled hyperglycaemia with a glucose level >240 mg/dL (>13.3 mmol/L)
* Impaired renal function, defined as estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 (moderate and severe renal impairment, modification of diet in renal disease (MDRD) formula)
* Acute coronary syndrome, stroke or transient ischemic attack (TIA) within 12 weeks prior to informed consent
* Indication of liver disease, defined by serum levels of either alanine transaminase (ALT), aspartate transaminase (AST), or alkaline phosphatase (ALP) above 3 x upper limit of normal (ULN)

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Japan (2):
  - 1245.35.002 Boehringer Ingelheim Investigational Site, Shinjyuku-ku, Tokyo
  - 1245.35.001 Boehringer Ingelheim Investigational Site, Suita-shi, Osaka

REFERENCES:
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Nishimura R, Tanaka Y, Koiwai K, Ishida K, Salsali A, Kaspers S, Kohler S, Lund SS. Effect of Empagliflozin on Free Fatty Acids and Ketone Bodies in Japanese Patients with Type 2 Diabetes Mellitus: A Randomized Controlled Trial. Adv Ther. 2019 Oct;36(10):2769-2782. doi: 10.1007/s12325-019-01045-x. Epub 2019 Aug 23. PMID 31444706
- [Derived] Nishimura R, Tanaka Y, Koiwai K, Inoue K, Hach T, Salsali A, Lund SS, Broedl UC. Effect of empagliflozin monotherapy on postprandial glucose and 24-hour glucose variability in Japanese patients with type 2 diabetes mellitus: a randomized, double-blind, placebo-controlled, 4-week study. Cardiovasc Diabetol. 2015 Jan 30;14:11. doi: 10.1186/s12933-014-0169-9. PMID 25633683

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablets matching empagliflozin 10 mg or 25 mg tablets
- Empagliflozin 10 mg: Empagliflozin 10 mg oral administration once daily
- Empagliflozin 25 mg: Empagliflozin 25mg oral administration once daily
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 21 | 20 | 19
Completed | 20 | 20 | 19
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: all patients treated with at least 1 dose of randomised study drug, and with a baseline AUC1-4h for plasma glucose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 21 | 20 | 19 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.8) | 64.8 (5.9) | 62.6 (7.8) | 62.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 13
  Male | 17 | 14 | 16 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in Area Under the Concentration-time Curve (AUC1-4h) for Postprandial Plasma Glucose From Baseline After 28 Days of Treatment
Description: The primary endpoint is the change in AUC1-4h for postprandial plasma glucose based on meal tolerance test from baseline after 28 days of treatment. Baseline refers to the last observation prior to administration of randomised study medication.
Time Frame: 1h, 1.5h, 2h, 2.5, 3h, 3.5h and 4h after drug administration at day -1 (baseline), and 1h, 1.5h, 2h, 2.5, 3h, 3.5h and 4h after drug administration at day 28
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg*h/dL
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 20 | 20 | 19
mg*h/dL | -18.07 (13.89) | -103.56 (14.24) | -122.94 (14.35)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 25 mg; Difference calculated as empa 25 mg minus placebo. The analyses will be performed sequentially compared with placebo from high dose of empagliflozin and the full significance level (5%) will be maintained by the hierarchical procedure; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment, number of previous antidiabetic medication, baseline renal function, baseline HbA1c and baseline AUC1-4h for plasma glucose; Mean Difference (Net) = -104.87, 95% CI 2-sided [-144.77 to -64.97], Standard Error of Mean 19.88
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 10 mg; Difference calculated as empa 10 mg minus placebo. The analyses will be performed sequentially compared with placebo from high dose of empagliflozin and the full significance level (5%) will be maintained by the hierarchical procedure; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -85.49, 95% CI 2-sided [-126.01 to -44.97], Standard Error of Mean 20.18

ADVERSE EVENTS:
Time Frame: between the first drug intake of study medication and 7 days after last drug intake of study medication, up to 35 days
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 1/21 | 2/20 | 3/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Empagliflozin 10 mg (N=20) | Empagliflozin 25 mg (N=19)
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Bartholinitis (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.